CLINICAL TRIAL: NCT04117841
Title: SLIP Registry - SCFE Longitudinal International Prospective Registry
Brief Title: SCFE Longitudinal International Prospective Registry
Acronym: SLIP
Status: Recruiting | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kishore Mulpuri, Principal Investigator, University of British Columbia
Other Study IDs: H15-03132
Record Dates: First submitted 2019-10-02; First posted 2019-10-07 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Slipped Capital Femoral Epiphyses; SCFE
MeSH Terms: conditions — Slipped Capital Femoral Epiphyses | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Arm I: Prospective from diagnosis: Patients have been enrolled and followed since diagnosis will be placed into Arm I.
  Interventions: Other: Observational
- Arm II: Prior treatment at centre: Patients who have received previous treatment and will continue to receive treatment at the participating center will be placed into Arm II.
  Interventions: Other: Observational
- Arm III: Prior treatment at outside centre: Patients who have received previous treatment at an outside center but are continuing treatment at a participating center will be placed into Arm III.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — All groups will undergo observational data collection. No interventions will be made to patient care.

SUMMARY:
Slipped Capital Femoral Epiphysis (SCFE) is the most common disorder of the adolescent hip and diagnosis and treatment of SCFE remain areas of controversy and investigation. The current issues relating to diagnosis stem from an inability to diagnose the condition early on, resulting in increased morbidity. Once diagnosed, there are multiple different options for surgical treatment, including in-situ pinning, and the Modified Dunn procedure. Research is ongoing to determine the parameters that should be considered when selecting a procedure to ensure an ideal outcome. In particular, there is a focus on investigating which treatment method may result in lower incidence of avascular necrosis of the femoral head and femoroacetabular impingement (FAI), two significant long term concerns associated with SCFE. Despite myriad published studies on SCFE, very few are prospective and most lack sufficient patient numbers for clinically meaningful comparative analysis. The aim of this study is to develop a multi-center, international prospective registry of patients with SCFE to facilitate the comprehensive examination of clinical, functional and radiographic outcomes of each treatment, in relation to specific parameters determined prior to intervention. The general registry will serve as a hypothesis-generating database of prospectively collected outcomes. In turn, this will facilitate the development of targeted, hypothesis-testing randomized controlled trials and observational studies that can be housed within the larger registry.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of SCFE
* Intend to receiving follow-up at participating centre
* Less than 18 years old at time of admission
* Adequate diagnostic information and radiographic imaging (for patients previously treated for SCFE)

Exclusion Criteria:

* No definitive diagnosis of SCFE
* Do not intend to receive follow-up at a participating centre
* Greater than 18 years old at time of admission
* Prior treatment for SCFE not appropriately documented
* Known or suspected underlying conditions (e.g., cerebral palsy, spina bifida, or osteogenesis imperfecta)

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who have been diagnosed with SCFE and receive follow-up at a participating centre will be included in the registry. Patients will be enrolled during one of their routine clinic appointments at one of the participating centers.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-05-30 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Development of a multi-centre, general, prospective SCFE registry, with follow-up to skeletal maturity | Until study completion in 2028
Comparison of the clinical, functional, and radiographic parameters related to SCFE in the context of treatment outcomes | Until study completion in 2028
Examination of the long-term outcome of prophylactically pinning the contralateral hip, specifically in regards to development of avascular necrosis | Until study completion in 2028
Determination of whether prophylactic fixation allows for preservation of hip morphology and function in the short and long term | Until study completion in 2028
Comparative analysis of surgical treatment outcomes, with particular regard to complications (avascular necrosis, femoroacetabular impingement (FAI), secondary surgeries) | Until study completion in 2028
Comparison of mild SCFE treatment with or without acute FAI treatment in regard to complication and short-term outcomes | Until study completion in 2028
Examination of timelines and results of diagnostic tests leading to the diagnosis of SCFE | Until study completion in 2028
Determination of the timeline for patients to return to full weight-bearing following treatment and to assess the level to which they return to activity | Until study completion in 2028

CONTACTS AND LOCATIONS:
Overall Officials: Kishore Mulpuri, FRCSC, Principal Investigator — Principal Investigator
Locations (1):
- British Columbia Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No